CLINICAL TRIAL: NCT04248101
Title: Comparison of Double Ligation and Topical Silver Nitrate for Treatment of Umbilical Granuloma in Children: A Randomized Control Trial
Brief Title: Double Ligation and Topical Silver Nitrate
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Rashid, Scholar MS Paediatric Surgery, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Umbilical Granuloma
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Umbilical Granuloma
Keywords: Double Ligation, Topical Silver Nitrate
MeSH Terms: interventions — Silver Nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): 88 cases of umbilical granulomas who were treated with double ligation
  Interventions: Procedure: Double Ligation
- Group 2 (Active Comparator): 88 cases of umbilical granulomas who were treated with topical silver nitrate
  Interventions: Drug: Topical Silver Nitrate

INTERVENTIONS:
Procedure: Double Ligation
  Arms: Group 1
Drug: Topical Silver Nitrate
  Arms: Group 2

SUMMARY:
To study and compare the efficacy and safety of Double Ligation and Topical Silver Nitrate Solution while treating children with Umbilical Granulomas

DETAILED DESCRIPTION:
The patients underwent one treatment option and then followed up for three weeks and the results noted in terms of success/failure and complications specific to each treatment option and analysed accordingly

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Umbilical Granuloma, less than 1 year age

Exclusion Criteria:

1. Patients who already had any treatment
2. Parents refused to give consent for enrollment
3. Patients lost in follow up

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Success/Failure of treatment | 3 weeks
  The effect of treatment was noted in a structured proforma on weekly basis for 3 weeks.
  Treatment was considered successful if, on local examination the granuloma disappeared completely and did not reappear during the follow up period.
  And if the granuloma did not disppear completely during the follow up period after double ligation or application of silver nitrate, treatment was considered to have failed.
  These variables were measured as frequency and percentages. The results were compared between the two groups using chi-square test. A significance level of <0.05 was considered significant.
Frequency of complications in both groups | 3 weeks
  The complications were also noted in the above mentioned proforma during the follow up period on weekly basis for 3 weeks.
  Complications relevant to the treatment i.e. infection, bleeding, chemical burns and skin discoloration were noted during local examination.
  These variables were measured as frequency and percentages. The results were compared between the two groups using chi-square test. A significance level of <0.05 was considered significant

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Akhtar, MS Paediatric Surgery, Study Director — Professor of Paediatric Surgery

IPD SHARING:
Plan to Share IPD: No